CLINICAL TRIAL: NCT00119054
Title: Effectiveness of Care Coordination in Managing Medically Complex Patients
Brief Title: Effectiveness of Home-Based Health Messaging for Patients With Hypertension and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: NRI 03-312
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2008-01

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Hypertension; Diabetes Mellitus; Telemedicine; Nursing Care
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: In Home Health Messaging Device

INTERVENTIONS:
Behavioral: In Home Health Messaging Device

SUMMARY:
Patients treated at Veterans Affairs (VA) medical centers are older and have multiple chronic conditions. Two of the most common conditions in the VA population are hypertension (HTN) and Type 2 diabetes (DM). Unfortunately, DM and HTN have few perceptible symptoms on a daily basis that motivate patients to comply with treatment recommendations and lifestyle changes. Thus, serious complications and long-term adverse outcomes are common in both of these conditions.

Home telehealth is a general term used to describe the delivery of health care services to the patient's home using audio, video, or other telecommunications technologies. Although home telehealth offers a number of theoretical advantages, few well-designed controlled clinical trials have been conducted to establish efficacy and cost benefit. Furthermore, projects to date have focused on special populations, e.g., heart failure or mental illnesses. Since home telehealth may hold the most promise for individuals dealing with multiple chronic illnesses, there is a need for population-based studies addressing the needs of patients in primary care settings.

Care coordination, as defined by the VHA Office of Care Coordination, is a process of assessment and ongoing monitoring of patients using home telehealth to proactively enable prevention, investigation, and treatment that enhances the health of patients and prevents unnecessary and inappropriate use of resources. Care coordination embeds technology into a care management process. This results in the right care, at the right time, in the right place.

DETAILED DESCRIPTION:
Patients treated at Veterans Affairs (VA) medical centers are older and have multiple chronic conditions. Two of the most common conditions in the VA population are hypertension (HTN) and Type 2 diabetes (DM). Unfortunately, DM and HTN have few perceptible symptoms on a daily basis that motivate patients to comply with treatment recommendations and lifestyle changes. Thus, serious complications and long-term adverse outcomes are common in both of these conditions.

Home telehealth is a general term used to describe the delivery of health care services to the patient's home using audio, video, or other telecommunications technologies. Although home telehealth offers a number of theoretical advantages, few well-designed controlled clinical trials have been conducted to establish efficacy and cost benefit. Furthermore, projects to date have focused on special populations, e.g., heart failure or mental illnesses. Since home telehealth may hold the most promise for individuals dealing with multiple chronic illnesses, there is a need for population-based studies addressing the needs of patients in primary care settings.

Care coordination, as defined by the VHA Office of Care Coordination, is a process of assessment and ongoing monitoring of patients using home telehealth to proactively enable prevention, investigation, and treatment that enhances the health of patients and prevents unnecessary and inappropriate use of resources. Care coordination embeds technology into a care management process. This results in the right care, at the right time, in the right place.The primary objective of the proposed study is to evaluate the efficacy of care coordination in improving outcomes in veterans with co-morbid DM and HTN, the two most common chronic conditions seen in VA Primary Care clinics. The specific aim is to compare outcomes of patients who receive the care coordination intervention to outcomes of patients who receive usual care. Three hypotheses will be tested: Compared to subjects who receive usual care, subjects who receive the care coordination intervention will have: 1) improved clinical measures [hemoglobin A1c (HbA1c) and systolic blood pressure (SBP)] at 6 and 12 months after study enrollment; 2) improved disease self-management (knowledge, self-efficacy, and adherence) at 6 and 12 months after study enrollment; and 3) improved quality of life and satisfaction with care at 6 and 12 months after study enrollment.Subjects wererecruited from VA Primary Care clinic rolls. 302 subjects were randomized to three groups: low-intensity monitoring plus nurse care management intervention (n=102); high-intensity monitoring plus nurse care management intervention (n=93); and usual care (n=107). In both intervention groups patients transmitted vital signs daily. In addition, the low intensity group answered two general health questions; the high intensity group responded to a complete range of questions focused on diabetes and hypertension, and received educational tips. The intervention groups participated in the protocol for 6 months following enrollment. Data were collected at baseline and at 6 and 12 months, including measures of clinical outcomes, quality of life, knowledge, adherence, self-efficacy, and satisfaction with care. In addition to these measures, data were collected to estimate the cost of the home telehealth intervention. Most subjects were male (98%) Caucasians (96%) with a mean age of 68 years (range 40-89 years).

ELIGIBILITY:
Inclusion Criteria:

Patients must obtain their primary care at the Iowa City VAMC and have been diagnosed with Diabetes Mellitus and hypertension. Must be cognitively intact and have a telephone line in the home.

Exclusion Criteria:

Patients with corrected vision worse than 20/40 or cognitive impairment (Mini-Mental Status Exam score of 17 or less) will not be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2005-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Blood Pressure and Hemaglobin A1c

SECONDARY OUTCOMES:
Knowledge Compliance Self-efficacy Quality of life Satisfaction with care

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie J. Wakefield, PhD RN, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

REFERENCES:
- [Result] Wakefield BJ, Holman JE, Ray A, Scherubel M, Adams MR, Hills SL, Rosenthal GE. Outcomes of a home telehealth intervention for patients with diabetes and hypertension. Telemed J E Health. 2012 Oct;18(8):575-9. doi: 10.1089/tmj.2011.0237. Epub 2012 Aug 8. PMID 22873700
- [Result] Wakefield BJ, Holman JE, Ray A, Scherubel M, Adams MR, Hillis SL, Rosenthal GE. Effectiveness of home telehealth in comorbid diabetes and hypertension: a randomized, controlled trial. Telemed J E Health. 2011 May;17(4):254-61. doi: 10.1089/tmj.2010.0176. Epub 2011 Apr 10. PMID 21476945
- [Result] Wakefield BJ, Holman JE, Ray A, Scherubel M. Patient perceptions of a remote monitoring intervention for chronic disease management. J Gerontol Nurs. 2011 Apr;37(4):16-20. doi: 10.3928/00989134-20110302-05. Epub 2011 Mar 16. PMID 21417194
- [Result] Young LB, Foster L, Silander A, Wakefield BJ. Home telehealth: patient satisfaction, program functions, and challenges for the care coordinator. J Gerontol Nurs. 2011 Nov;37(11):38-46. doi: 10.3928/00989134-20110706-02. Epub 2011 Jul 15. PMID 21761815
- [Result] Wakefield BJ, Scherubel M, Ray A, Holman JE. Nursing interventions in a telemonitoring program. Telemed J E Health. 2013 Mar;19(3):160-5. doi: 10.1089/tmj.2012.0098. Epub 2013 Jan 28. PMID 23356382
- [Result] Gardner SE, Hillis SL, Frantz RA. Clinical signs of infection in diabetic foot ulcers with high microbial load. Biol Res Nurs. 2009 Oct;11(2):119-28. doi: 10.1177/1099800408326169. PMID 19147524
- [Result] Boren SA, Wakefield BJ, Dohrmann M. Chronic heart failure consumer information: an exploratory study. AMIA Annu Symp Proc. 2008 Nov 6:884. PMID 18998896
- [Result] Wakefield BJ, Mentes J, Holman JE, Culp K. Postadmission dehydration: risk factors, indicators, and outcomes. Rehabil Nurs. 2009 Sep-Oct;34(5):209-16. doi: 10.1002/j.2048-7940.2009.tb00281.x. PMID 19772119
- [Result] Rantz MJ, Skubic M, Alexander G, Popescu M, Aud MA, Wakefield BJ, Koopman RJ, Miller SJ. Developing a comprehensive electronic health record to enhance nursing care coordination, use of technology, and research. J Gerontol Nurs. 2010 Jan;36(1):13-7. doi: 10.3928/00989134-20091204-02. Epub 2010 Jan 12. PMID 20047248